CLINICAL TRIAL: NCT03192774
Title: A Prospective Follow-up Assessment of Transcatheter Aortic Valve Implantation in Bad Segeberg
Brief Title: The Prospective Segeberg TAVI Registry
Acronym: POST-TAVI
Status: Recruiting | Type: Observational
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SK 109 -- 168/11
Record Dates: First submitted 2017-06-18; First posted 2017-06-20 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Interventional replacement of the aortic valve

SUMMARY:
A single center registry including all patients treated with TAVI at the Heart Center, Bad Segeberg, Germany

DETAILED DESCRIPTION:
A prospective single center registry including all patients treated with transcatheter aortic valve implantation (TAVI) at the Heart Center, Bad Segeberg, Germany. Patients undergo a routine clinical and echocardiographic follow-up schedule, including a long-term follow-up plan beyond 5 years to assess valve durability.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with TAVI

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers patient population treated with TAVI.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 10 years
  Cardiovascular and not cardiovascular death

SECONDARY OUTCOMES:
Structural valve deterioration | Up to 10 years
  Transprosthetic mean pressure gradient ≥40 mmHg and/or ≥20 mmHg rise from baseline OR severe intraprosthetic aortic regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Gert Richardt, MD, Study Chair — Heart Center, Segeberger Kliniken; Mohamed Abdel-Wahab, MD, Principal Investigator — Heart Center, Segeberger Kliniken
Locations (1):
- Heart Center, Segeberger Kliniken, Bad Segeberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amoey D, Samy M, Elbasha K, Alali A, Landt M, Kurniadi A, Nef H, Tolg R, Richardt G, Mankerious N. Predictors and Outcomes of Inappropriate Dosing of Direct Oral Anticoagulants in Patients Receiving Transcatheter Aortic Valve Implantation. Cardiol Ther. 2024 Dec;13(4):761-773. doi: 10.1007/s40119-024-00387-0. Epub 2024 Nov 4. PMID 39495243
- [Derived] Samy M, Landt M, Mankerious N, Kurniadi A, Alotaibi S, Toelg R, Abdel-Wahab M, Nef H, Allali A, Richardt G, Elbasha K. ProGlide-AngioSeal versus ProGlide-FemoSeal for vascular access hemostasis posttranscatheter aortic valve implantation. Catheter Cardiovasc Interv. 2024 Nov;104(6):1251-1259. doi: 10.1002/ccd.31259. Epub 2024 Oct 8. PMID 39378384
- [Derived] Alotaibi S, Elbasha K, Landt M, Kaur J, Kurniadi A, Abdel-Wahab M, Toelg R, Richardt G, Allali A. Prognostic Value of HFA-PEFF Score in Patients Undergoing Transcatheter Aortic Valve Implantation. Cureus. 2022 Jul 22;14(7):e27152. doi: 10.7759/cureus.27152. eCollection 2022 Jul. PMID 36017287
- [Derived] Abdelghani M, Mankerious N, Landt M, Toelg R, Abdel-Wahab M, Richardt G. Transcatheter Aortic Valve Implantation With the Third Generation Balloon-Expandable Bioprosthesis in Patients With Severe Landing Zone Calcium. Am J Cardiol. 2020 Mar 15;125(6):931-940. doi: 10.1016/j.amjcard.2019.12.022. Epub 2019 Dec 27. PMID 31959428